CLINICAL TRIAL: NCT04676867
Title: A Double-blind, Placebo-controlled, Phase 2a Proof-of-concept Trial of Dalcetrapib in Patients With Confirmed Mild to Moderate COVID-19
Brief Title: Effect of Dalcetrapib in Patients With Confirmed Mild to Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DalCor Pharmaceuticals (Industry)
Collaborators: The Montreal Health Innovations Coordinating Center (MHICC) (Other); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAL-401
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Results first posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID-19; Coronavirus disease; Dalcetrapib
MeSH Terms: conditions — COVID-19 | interventions — dalcetrapib

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blind, multicenter, Phase 2a proof-of-concept study in outpatients with confirmed, mild to moderate, symptomatic COVID-19.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 900 mg dose (Active Comparator): Patients will receive Dalcetrapib 900 mg for 10 days
  Interventions: Drug: Dalcetrapib
- 1800 mg dose (Active Comparator): Patients will receive Dalcetrapib 1800 mg for 10 days
  Interventions: Drug: Dalcetrapib
- 3600 mg dose (Active Comparator): Patients will receive Dalcetrapib 3600 mg for 10 days
  Interventions: Drug: Dalcetrapib
- Placebo tablets (Placebo Comparator): Patients will receive Placebo for 10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dalcetrapib — Dalcetrapib 300 mg Film-Coated Tablets
  Arms: 1800 mg dose; 3600 mg dose; 900 mg dose
Other: Placebo — Placebo Tablets
  Arms: Placebo tablets

SUMMARY:
This study is a placebo-controlled, Phase 2a proof-of-concept clinical study which will evaluate efficacy and safety of dalcetrapib in outpatients patients with mild to moderate, symptomatic, confirmed COVID 19.

ELIGIBILITY:
Inclusion Criteria:

* Patients must satisfy all of the following criteria unless otherwise stated:

  1. Willing and able to provide informed consent
  2. Male or female patients > 18 years of age on the day of informed consent
  3. Have received a confirmed diagnosis of COVID-19 (positive for SARS CoV 2), as assessed by PCR or point-of-care within 72 hours of first dose on Day 1
  4. Have mild to moderate signs or symptoms of COVID-19 with onset within 5 days of first dose on Day 1, at least two of the following symptoms:

     * stuffy or runny nose
     * sore throat
     * shortness of breath
     * cough
     * fatigue
     * myalgia
     * headache
     * chills or shivering
     * feeling hot or feverish
     * nausea
     * vomiting
     * diarrhea
     * anosmia
     * ageusia
  5. Outpatient with COVID-19 disease (not requiring oxygen therapy [WHO COVID-19 Clinical Improvement Ordinal Scale, score of 3])
  6. Patient is aware of the investigational nature of this study and willing to comply with protocol treatments, blood tests, and other evaluations listed in the informed consent form (ICF).

Exclusion Criteria:

* Patients will be excluded from the study if they satisfy any of the following criteria unless otherwise stated:

  1. Females who are pregnant (negative pregnancy test required for all women of child bearing potential at Screening) or breast-feeding
  2. Male patients and women of childbearing potential (women who are not surgically sterile or postmenopausal defined as amenorrhea for >12 months) who are not using at least one protocol specified method of contraception
  3. Severe COVID-19 disease as defined by the WHO COVID-19 Clinical Improvement Ordinal Scale, scores of 5 (non invasive ventilation or high-flow oxygen), 6 (intubation and mechanical ventilation), or 7 (ventilation + additional organ support pressors, renal replacement therapy [RRT], extracorporeal membrane oxygenation [ECMO])
  4. Expected survival less than 72 hours
  5. Peripheral capillary oxygen saturation (SpO2) <90% while breathing room air
  6. Treatment with other drugs thought to possibly have activity against SARS CoV 2 infection like remdesivir, favipiravir, within 7 days prior to enrollment or concurrently
  7. History of abuse of drugs or alcohol that could interfere with adherence to study requirements as judged by the Investigator
  8. Use of any other concurrent investigational drugs while participating in the present study
  9. Patient requires frequent or prolonged use of systemic corticosteroids (≥20 mg of prednisone/day or equivalent for >4 weeks) or other immunosuppressive drugs (e.g., for organ transplantation or autoimmune conditions)
  10. Known renal disease with an estimated glomerular filtration rate (eGFR) <50 mL/min based on local laboratory results
  11. Patients with clinically apparent liver disease, e.g., jaundice, cholestasis, hepatic synthetic impairment, or active hepatitis
  12. Alanine transaminase (ALT) or aspartate transaminase (AST) >3 × upper limit of normal (ULN) or alkaline phosphatase or bilirubin levels > 2 × ULN based on local laboratory results
  13. Co administration of clinical doses of orlistat with dalcetrapib
  14. Inability to swallow oral medications or a gastrointestinal disorder with diarrhea (e.g., Crohn's disease) or malabsorption at Screening
  15. Any other clinically significant medical condition or laboratory abnormality that, in the opinion of the Investigator, would jeopardize the safety of the patient or potentially impact patient compliance or the safety/efficacy observations in the study
  16. History of an allergic reaction or hypersensitivity to the study drug or any component of the study drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kallend, Study Director — DalCor Pharmaceuticals
Locations (1):
- Institut de Cardiologie de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Department of Health and Human Services, Determination of a Public Health Emergency and Declaration that Circumstances Exist Justifying Authorizations Pursuant to Section 564(b) of the Federal Food, Drug, and Cosmetic Act, 21 U.S.C. § 360bbb-3. February 4, 2020.
- [Background] Schwartz GG, Olsson AG, Abt M, Ballantyne CM, Barter PJ, Brumm J, Chaitman BR, Holme IM, Kallend D, Leiter LA, Leitersdorf E, McMurray JJ, Mundl H, Nicholls SJ, Shah PK, Tardif JC, Wright RS; dal-OUTCOMES Investigators. Effects of dalcetrapib in patients with a recent acute coronary syndrome. N Engl J Med. 2012 Nov 29;367(22):2089-99. doi: 10.1056/NEJMoa1206797. Epub 2012 Nov 5. PMID 23126252
- [Background] Dai W, Zhang B, Jiang XM, Su H, Li J, Zhao Y, Xie X, Jin Z, Peng J, Liu F, Li C, Li Y, Bai F, Wang H, Cheng X, Cen X, Hu S, Yang X, Wang J, Liu X, Xiao G, Jiang H, Rao Z, Zhang LK, Xu Y, Yang H, Liu H. Structure-based design of antiviral drug candidates targeting the SARS-CoV-2 main protease. Science. 2020 Jun 19;368(6497):1331-1335. doi: 10.1126/science.abb4489. Epub 2020 Apr 22. PMID 32321856
- See also: World Health Organization. WHO Coronavirus Disease (COVID-19) Dashboard. — https://covid19.who.int/?gclid=CjwKCAjwm_P5BRAhEiwAwRzSO9jpEwPeoHR8NmLUmBMkH5BdQEdGyjVJa5ktZh6WxXPcKP3RaC2M_BoCO-UQAvD_BwE

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 227 subjects signed informed consent, 225 of whom were randomized to treatment (2 subjects were not randomized). Of these 225 randomized subjects, 17 subjects did not take any study medication (causes: failed screening criteria, lost to follow-up, or withdrew consent) and were excluded from all analyses. A total of 208 subjects (92.5%) entered the trial and received at least one dose of study medication.
Groups:
- Placebo Tablets: Participants received twelve dalcetrapib placebo tablets orally daily for 10 days.
  Placebo: Dalcetrapib matching placebo tablets
- 900 mg Dose: Participants received dalcetrapib 900 mg (three 300 mg tablets) and 9 placebo tablets orally daily for 10 days
  Dalcetrapib: Dalcetrapib 300 mg film-coated tablets Placebo: Dalcetrapib matching placebo tablets
- 1800 mg Dose: Participants received dalcetrapib 1800 mg (six 300 mg tablets) and six placebo tablets orally daily for 10 days
  Dalcetrapib: Dalcetrapib 300 mg film-coated tablets Placebo: Dalcetrapib matching placebo tablets
- 3600 mg Dose: Participants received dalcetrapib 900 mg (twelve 300 mg tablets) orally daily for 10 days
  Dalcetrapib: Dalcetrapib 300 mg film-coated tablets Placebo: Dalcetrapib matching placebo tablets
Period: Overall Study
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Started | 56 (Medication never taken n=3) | 56 (Medication never taken n=1) | 56 (Medication never taken n=8) | 57 (Medication never taken n=5)
Entered Study and Received at Least 1 Dose of Study Medication | 53 | 55 | 48 | 52
Completed | 53 | 54 | 45 | 51
Not Completed | 3 | 2 | 11 | 6
Not completed — Screen failure | 0 | 0 | 6 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 4 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 225 randomized subjects, a total of 208 subjects received at least one dose of study medication, for which baseline data are presented here. The overall number of baseline participants in each arm reflects the number of subjects who took at least one dose of study medication in each arm, not the total number randomized in each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose | Total
Number analyzed (Participants) | 53 | 55 | 48 | 52 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (13.2) | 46.7 (10.4) | 42.5 (12.0) | 46.5 (11.0) | 44.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 19 | 28 | 115
  Male | 19 | 21 | 29 | 24 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 1 | 7
  Not Hispanic or Latino | 51 | 53 | 46 | 50 | 200
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 53 | 53 | 45 | 51 | 202
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 53 | 55 | 48 | 52 | 208
Smoking status [Count of Participants; unit: Participants]
  Never smoker | 28 | 33 | 29 | 25 | 115
  Current smoker | 8 | 4 | 7 | 6 | 25
  Former smoker | 17 | 18 | 12 | 21 | 68

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Clinical Resolution of Symptoms of COVID-19 (Excluding Cough, Sense of Smell and Taste) in Subjects With Confirmed, Mild to Moderate, Symptomatic COVID-19 Treatment With Dalcetrapib
Description: Sustained clinical resolution is defined as occurring when no key COVID-19 related symptom has a score higher than 1 over a 72-hour period (as documented using an electronic patient-reported outcome [ePRO] instrument), except for sense of smell and taste where the score should be 0 over a 72-hour period. The time to resolution was taken as the time from randomization until the first day of the last 72-hour period where the patient met the definition of resolution within 28 days. Patients who did not meet the definition of resolution 28 days after randomization were considered not resolved.
  The scale is "Assessment of 14 Common COVID-19-Related Symptoms: Items and Response" from the Food and Drug Administration (FDA). The symptoms are scored as on a scale of 0 to 3 for 12 of the symptoms where 0 is none and on a scale of 0 to 2 for the two other symptoms where 0 is "as usual". A higher score is a worse outcome.
Time Frame: 28 days
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
days | 9.0 [8.0 to 14.0] | 9.0 [8.0 to 10.0] | 9.5 [8.0 to 14.0] | 10.0 [9.0 to 11.0]
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Log Rank

2. Secondary Outcome: Change From Baseline in log10 Viral Load (Saliva)
Description: Log10 viral load, as assessed using the saliva, was summarized by treatment group using descriptive statistics (N, mean, median, standard deviation, minimum, and maximum) for each visit as well as for changes from baseline where an 80% CI were also presented. A repeated ANCOVA model was used for the data shown below, showing the mean changes from baseline to study visits (Day 3, Day 5, Day 10, and Day 28/EOS) in log10 viral load including treatment groups by study visit interaction, baseline value of log10 viral load and baseline value of log10 viral load by study visit interaction.
Time Frame: Screening/Baseline (Day -2 to Day -1), Day 3, Day 5, Day 10, and Day 28/End of Study (EOS)
Measure: Mean (80% Confidence Interval); unit: log10 viral titers
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
log10 viral titers
  Day 3 | -0.77 [-1.04 to -0.49] | -0.79 [-1.04 to -0.54] | -0.61 [-0.89 to -0.32] | -0.79 [-1.07 to -0.51]
  Day 5 | -1.45 [-1.72 to -1.18] | -1.50 [-1.76 to -1.25] | -1.45 [-1.73 to -1.17] | -1.27 [-1.55 to -0.99]
  Day 10 | -3.43 [-3.79 to -3.08] | -3.24 [-3.55 to -2.92] | -3.01 [-3.38 to -2.65] | -3.23 [-3.61 to -2.85]
  Day 28/End of Study | -5.16 [-5.40 to -4.91] | -4.96 [-5.20 to -4.72] | -5.30 [-5.57 to -5.03] | -5.16 [-5.42 to -4.90]
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, ANCOVA

3. Secondary Outcome: Change From Baseline in log10 Viral Load (Nasal Swab)
Description: Log10 viral load, as assessed using the nasal swab, was summarized by treatment group using descriptive statistics (N, mean, median, standard deviation, minimum, and maximum) for each visit as well as for changes from baseline where an 80% CI were also presented. A repeated ANCOVA model was used for the data shown below, showing the mean changes from baseline to study visits (Day 3, Day 5, Day 10, and Day 28/EOS) in log10 viral load including treatment groups by study visit interaction, baseline value of log10 viral load and baseline value of log10 viral load by study visit interaction.
Time Frame: Screening/Baseline (Day -2 to Day -1), Day 3, Day 5, Day 10, and Day 28/End of Study (EOS)
Measure: Mean (80% Confidence Interval); unit: log10 viral titers
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
log10 viral titers
  Day 3 | -0.94 [-1.18 to -0.71] | -1.17 [-1.39 to -0.94] | -0.84 [-1.09 to -0.60] | -0.92 [-1.17 to -0.68]
  Day 5 | -1.87 [-2.15 to -1.60] | -2.25 [-2.53 to -1.98] | -1.47 [-1.76 to -1.17] | -2.00 [-2.29 to -1.71]
  Day 10 | -4.76 [-5.08 to -4.45] | -4.42 [-4.72 to -4.11] | -3.87 [-4.22 to -3.52] | -4.23 [-4.59 to -3.87]
  Day 28/End of Study | -6.24 [-6.32 to -6.15] | -6.29 [-6.38 to -6.21] | -6.26 [-6.36 to -6.17] | -6.34 [-6.43 to -6.25]
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, ANCOVA

4. Secondary Outcome: Time to Sustained Complete Clinical Resolution of Symptoms in Subjects With Confirmed, Mild to Moderate, Symptomatic COVID-19 Treatment With Dalcetrapib
Description: Sustained clinical resolution is defined as occurring when no key COVID-19 related symptom has a score higher than 1 over a 72-hour period (as documented using an electronic patient-reported outcome [ePRO] instrument). The time to resolution was taken as the time from randomization until the first day of the last 72-hour period where the patient met the definition of resolution within 28 days. Patients who did not meet the definition of resolution 28 days after randomization were considered not resolved.
  The scale is "Assessment of 14 Common COVID-19-Related Symptoms: Items and Response" from the Food and Drug Administration (FDA). The symptoms are scored as on a scale of 0 to 3 for 12 of the symptoms where 0 is none and on a scale of 0 to 2 for the two other symptoms where 0 is "as usual". A higher score is a worse outcome.
Time Frame: 28 days
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
days | 28.0 [16.0 to 28.0] | 28.0 [15.0 to 28.0] | 28.0 [28.0 to 29.0] | 28.0 [28.0 to 28.0]
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Log Rank

5. Secondary Outcome: Viral Clearance Using Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV-2) Polymerase Chain Reaction (PCR)
Description: Viral clearance based on polymerase chain reaction (PCR) test for Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV-2) using nasal swab and saliva samples was performed on the intention-to-treat (ITT) population. Viral clearance was summarized by treatment group using Kaplan-Meier methods. Median and associated 80% confidence interval (CI) was presented. The number and percentage of patients who did not show viral clearance, did show viral clearance, and patients censored were presented.
Time Frame: Day 1 to Day 28
Population: Two subjects were deleted from this analysis as the samples were deemed unreliable by the study site. One subject had no saliva samples analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 54 | 48 | 50
Participants
  Viral Clearance (saliva): Yes | 12 | 10 | 9 | 14
  Viral Clearance (saliva): No | 41 | 44 | 39 | 36
  Viral Clearance (nasal swab): Yes | 25 | 22 | 12 | 14
  Viral Clearance (nasal swab): No | 28 | 32 | 36 | 36
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Log Rank

6. Secondary Outcome: Time to Complete Clinical Resolution (Excluding Cough, Sense of Smell and Taste) Defined in the Same Way as the Primary Endpoint, But Considering That All Symptoms Must Resolve to a Score of 0 for 72 Hours
Description: Complete clinical resolution is defined as occurring when no key COVID-19 related symptom (excluding cough, sense of smell and taste) has a score higher than 0 over a 72-hour period. The time to resolution was taken as the time from randomization until the first day of the last 72 hour period where the patient met the definition of resolution within 28 days. Patients who did not meet the definition of resolution 28 days after randomization were considered not resolved.
  The scale is "Assessment of 14 Common COVID-19-Related Symptoms: Items and Response" was used. The symptoms are scored as on a scale of 0 to 3 for 12 of the symptoms where 0 is none and on a scale of 0 to 2 for the two other symptoms where 0 is "as usual". A higher score is a worse outcome.
Time Frame: 28 days
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
days | 28.0 [28.0 to 29.0] | 28.0 [28.0 to 28.0] | 28.0 [28.0 to 29.0] | 28.0 [28.0 to 29.0]
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Log Rank

7. Secondary Outcome: Time to Complete Clinical Resolution
Description: Sustained clinical resolution is defined as occurring when no key COVID-19 related symptom has a score higher than 0 over a 72-hour period. The time to resolution was taken as the time from randomization until the first day of the last 72 hour period where the patient met the definition of resolution within 28 days. Patients who did not meet the definition of resolution 28 days after randomization were considered not resolved.
  The scale is "Assessment of 14 Common COVID-19-Related Symptoms: Items and Response" was used. The symptoms are scored as on a scale of 0 to 3 for 12 of the symptoms where 0 is none and on a scale of 0 to 2 for the two other symptoms where 0 is "as usual". A higher score is a worse outcome.
  Resolution must have occurred within 28 days. Time of resolution of 29 days was imputed in censored subjects.
Time Frame: 28 days
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
days | 29.0 [28.0 to 29.0] | 28.0 [28.0 to 29.0] | 29.0 [28.0 to 29.0] | 28.5 [28.0 to 29.0]
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Log Rank

8. Secondary Outcome: Change From Baseline in Coronavirus Disease of 2019 (COVID-19) Total Symptom Severity Score Collected at All Time Points
Description: COVID-19 total symptom severity score was summarized by treatment group using descriptive statistics (N, mean, median, standard deviation, minimum, and maximum) for each visit as well as for changes from baseline where an 80% confidence interval (CI) was also presented. Mean changes from baseline were analyzed using a repeated measures ANCOVA model.
  The scale is "Assessment of 14 Common COVID-19-Related Symptoms: Items and Response" from the Food and Drug Administration (FDA) document "Assessing COVID-19-Related Symptoms in Outpatient Adult and Adolescent Subjects in Clinical Trials of Drugs and Biological Products for COVID-19 Prevention or Treatment Guidance for Industry". Symptoms are scored as on a scale of 0 to 3 for 12 the symptoms and on a scale of 0 to 2 for two symptoms. The sum of all 14 symptom scores is reported, where 0 is the minimum and 40 is the maximum. A higher score is a worse outcome.
Time Frame: Baseline, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 14 (follow-up visit 1), and Day 28 (end of study / follow-up visit 2)
Population: The number of subjects is different at baseline and at post-baseline visits. The difference in means is therefore not the same as the mean of the differences. The analysis has been conducted on the mean of the differences and the analysis of the change from baseline to Day X is based on subjects who had data at both baseline and Day X visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
score on a scale
  Baseline | 10.70 (4.98) | 11.11 (4.34) | 10.88 (4.63) | 9.02 (3.92)
  Day 2: number analyzed (Participants) | 53 | 54 | 47 | 49
  Day 2 | 10.30 (5.35) | 10.76 (4.58) | 11.55 (4.29) | 11.39 (5.06)
  Change from baseline to Day 2: number analyzed (Participants) | 53 | 54 | 47 | 49
  Change from baseline to Day 2 | -0.40 (3.85) | -0.39 (3.52) | 0.68 (3.65) | 2.35 (3.90)
  Day 3: number analyzed (Participants) | 53 | 55 | 47 | 49
  Day 3 | 8.85 (4.79) | 9.42 (4.53) | 10.57 (5.04) | 10.12 (5.40)
  Change from baseline to Day 3: number analyzed (Participants) | 53 | 55 | 47 | 49
  Change from baseline to Day 3 | -1.85 (3.78) | -1.69 (3.80) | -0.38 (4.46) | 1.08 (4.71)
  Day 4: number analyzed (Participants) | 50 | 53 | 48 | 47
  Day 4 | 8.24 (5.13) | 9.60 (5.09) | 10.75 (5.87) | 9.34 (5.39)
  Change from baseline to Day 4: number analyzed (Participants) | 50 | 53 | 48 | 47
  Change from baseline to Day 4 | -2.54 (5.04) | -1.55 (4.73) | -0.13 (5.27) | 0.23 (5.03)
  Day 5: number analyzed (Participants) | 52 | 54 | 48 | 45
  Day 5 | 7.90 (4.97) | 8.89 (5.56) | 9.29 (4.78) | 8.36 (4.50)
  Change from baseline to Day 5: number analyzed (Participants) | 52 | 54 | 48 | 45
  Change from baseline to Day 5 | -2.79 (4.64) | -2.26 (4.98) | -1.58 (6.03) | -0.56 (4.47)
  Day 6: number analyzed (Participants) | 51 | 53 | 43 | 45
  Day 6 | 6.98 (5.09) | 7.94 (5.44) | 8.09 (4.86) | 8.24 (6.23)
  Change from baseline to Day 6: number analyzed (Participants) | 51 | 53 | 43 | 45
  Change from baseline to Day 6 | -3.67 (5.57) | -3.23 (5.32) | -2.44 (5.56) | -0.71 (5.61)
  Day 7: number analyzed (Participants) | 51 | 51 | 46 | 43
  Day 7 | 6.0 (5.5) | 5.75 (3.94) | 8.39 (6.49) | 6.91 (4.57)
  Change from baseline to Day 7: number analyzed (Participants) | 51 | 51 | 46 | 43
  Change from baseline to Day 7 | -4.65 (5.77) | -5.29 (4.85) | -2.24 (7.20) | -2.02 (4.58)
  Day 8: number analyzed (Participants) | 48 | 50 | 45 | 46
  Day 8 | 5.06 (4.14) | 5.82 (4.13) | 7.02 (6.25) | 5.50 (4.03)
  Change from baseline to Day 8: number analyzed (Participants) | 48 | 50 | 45 | 46
  Change from baseline to Day 8 | -5.48 (5.34) | -5.38 (4.76) | -3.64 (6.88) | -3.48 (4.18)
  Day 9: number analyzed (Participants) | 48 | 50 | 42 | 41
  Day 9 | 4.44 (3.76) | 5.22 (4.34) | 6.86 (6.45) | 4.90 (2.80)
  Change from baseline to Day 9: number analyzed (Participants) | 48 | 50 | 42 | 41
  Change from baseline to Day 9 | -6.10 (5.88) | -6.20 (4.75) | -4.00 (7.58) | -3.95 (4.39)
  Day 10: number analyzed (Participants) | 49 | 52 | 41 | 44
  Day 10 | 3.90 (3.62) | 4.37 (3.79) | 5.85 (6.67) | 4.00 (2.96)
  Change from baseline to Day 10: number analyzed (Participants) | 49 | 52 | 41 | 44
  Change from baseline to Day 10 | -6.67 (5.41) | -6.96 (4.25) | -4.59 (7.56) | -4.77 (4.36)
  Follow-up visit 1 (Day 14): number analyzed (Participants) | 50 | 51 | 44 | 43
  Follow-up visit 1 (Day 14) | 3.22 (3.72) | 3.39 (3.23) | 4.23 (6.19) | 3.40 (3.58)
  Change from baseline to follow-up visit 1: number analyzed (Participants) | 50 | 51 | 44 | 43
  Change from baseline to follow-up visit 1 | -7.42 (5.74) | -7.90 (4.35) | -6.59 (7.24) | 5.21 (4.95)
  Follow-up visit 2 (Day 28/End of Study): number analyzed (Participants) | 50 | 53 | 45 | 48
  Follow-up visit 2 (Day 28/End of Study) | 1.84 (2.49) | 2.23 (2.85) | 2.89 (6.20) | 1.75 (2.05)
  Change from baseline to follow-up visit 2: number analyzed (Participants) | 50 | 53 | 45 | 48
  Change from baseline to follow-up visit 2 | -8.96 (5.14) | -9.02 (4.26) | -7.78 (7.12) | -7.17 (4.74)
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, ANCOVA

9. Secondary Outcome: Scoring of World Health Organization (WHO) Clinical Outcome Scale (9-point Scale) at Screening, Days 1, 3, 5, End of Treatment (Day 10), Follow-Up Visit (Day 14), and Day 28
Description: The number and percentage of patients for each WHO clinical outcome score was summarized. Scores were compared using the Mann-Whitney-Wilcoxon test.
  This scale is called the "WHO Clinical Outcome Scale". It is scored from 0 to 9 where 9 is the most severe disease presentation. A higher score is a worse outcome.
Time Frame: Screening (Day -2 to Day -1), Days 1, 3, 5, End of Treatment (Day 10), Follow-Up Visit (Day 14), and Day 28
Population: Not all subjects completed the trial. World Health Organization Clinical Outcome Scores were not collected for withdrawn subjects beyond their withdrawal date.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
Participants
  Screening: WHO Clinical Outcome Scale Score 0 | 0 | 0 | 0 | 0
  Screening: WHO Clinical Outcome Scale Score 1 | 18 | 15 | 19 | 23
  Screening: WHO Clinical Outcome Scale Score 2 | 35 | 40 | 29 | 29
  Screening: WHO Clinical Outcome Scale Score 3 | 0 | 0 | 0 | 0
  Screening: WHO Clinical Outcome Scale Score 4 | 0 | 0 | 0 | 0
  Screening: WHO Clinical Outcome Scale Score 5 | 0 | 0 | 0 | 0
  Screening: WHO Clinical Outcome Scale Score 6 | 0 | 0 | 0 | 0
  Screening: WHO Clinical Outcome Scale Score 7 | 0 | 0 | 0 | 0
  Screening: WHO Clinical Outcome Scale Score 8 | 0 | 0 | 0 | 0
  Day 1: WHO Clinical Outcome Scale Score 0 | 0 | 0 | 0 | 0
  Day 1: WHO Clinical Outcome Scale Score 1 | 15 | 13 | 17 | 18
  Day 1: WHO Clinical Outcome Scale Score 2 | 38 | 42 | 31 | 34
  Day 1: WHO Clinical Outcome Scale Score 3 | 0 | 0 | 0 | 0
  Day 1: WHO Clinical Outcome Scale Score 4 | 0 | 0 | 0 | 0
  Day 1: WHO Clinical Outcome Scale Score 5 | 0 | 0 | 0 | 0
  Day 1: WHO Clinical Outcome Scale Score 6 | 0 | 0 | 0 | 0
  Day 1: WHO Clinical Outcome Scale Score 7 | 0 | 0 | 0 | 0
  Day 1: WHO Clinical Outcome Scale Score 8 | 0 | 0 | 0 | 0
  Day 3: number analyzed (Participants) | 53 | 54 | 47 | 44
  Day 3: WHO Clinical Outcome Scale Score 0 | 0 | 0 | 0 | 0
  Day 3: WHO Clinical Outcome Scale Score 1 | 18 | 16 | 15 | 19
  Day 3: WHO Clinical Outcome Scale Score 2 | 35 | 38 | 32 | 25
  Day 3: WHO Clinical Outcome Scale Score 3 | 0 | 0 | 0 | 0
  Day 3: WHO Clinical Outcome Scale Score 4 | 0 | 0 | 0 | 0
  Day 3: WHO Clinical Outcome Scale Score 5 | 0 | 0 | 0 | 0
  Day 3: WHO Clinical Outcome Scale Score 6 | 0 | 0 | 0 | 0
  Day 3: WHO Clinical Outcome Scale Score 7 | 0 | 0 | 0 | 0
  Day 3: WHO Clinical Outcome Scale Score 8 | 0 | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 51 | 53 | 42 | 46
  Day 5: WHO Clinical Outcome Scale Score 0 | 0 | 0 | 1 | 0
  Day 5: WHO Clinical Outcome Scale Score 1 | 17 | 21 | 12 | 19
  Day 5: WHO Clinical Outcome Scale Score 2 | 34 | 31 | 29 | 27
  Day 5: WHO Clinical Outcome Scale Score 3 | 0 | 0 | 0 | 0
  Day 5: WHO Clinical Outcome Scale Score 4 | 0 | 1 | 0 | 0
  Day 5: WHO Clinical Outcome Scale Score 5 | 0 | 0 | 0 | 0
  Day 5: WHO Clinical Outcome Scale Score 6 | 0 | 0 | 0 | 0
  Day 5: WHO Clinical Outcome Scale Score 7 | 0 | 0 | 0 | 0
  Day 5: WHO Clinical Outcome Scale Score 8 | 0 | 0 | 0 | 0
  End of Treatment (Day 10): number analyzed (Participants) | 52 | 54 | 47 | 50
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 0 | 3 | 5 | 5 | 1
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 1 | 29 | 27 | 19 | 18
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 2 | 19 | 20 | 22 | 31
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 3 | 1 | 0 | 1 | 0
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 4 | 0 | 2 | 0 | 0
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 5 | 0 | 0 | 0 | 0
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 6 | 0 | 0 | 0 | 0
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 7 | 0 | 0 | 0 | 0
  End of Treatment (Day 10): WHO Clinical Outcome Scale Score 8 | 0 | 0 | 0 | 0
  Follow-up visit 1 (Day 14): number analyzed (Participants) | 52 | 54 | 44 | 48
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 0 | 10 | 14 | 12 | 13
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 1 | 31 | 21 | 23 | 24
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 2 | 11 | 18 | 8 | 11
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 3 | 0 | 1 | 0 | 0
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 4 | 0 | 0 | 0 | 0
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 5 | 0 | 0 | 0 | 0
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 6 | 0 | 0 | 0 | 0
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 7 | 0 | 0 | 1 | 0
  Follow-up visit 1 (Day 14): WHO Clinical Outcome Scale Score 8 | 0 | 0 | 0 | 0
  Follow-up visit 2 (Day 28/End Of Study): number analyzed (Participants) | 53 | 54 | 46 | 51
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 0 | 28 | 21 | 19 | 19
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 1 | 20 | 21 | 21 | 24
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 2 | 5 | 12 | 5 | 8
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 3 | 0 | 0 | 0 | 0
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 4 | 0 | 0 | 0 | 0
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 5 | 0 | 0 | 0 | 0
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 6 | 0 | 0 | 0 | 0
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 7 | 0 | 0 | 0 | 0
  Follow-up visit 2 (Day 28/End Of Study): WHO Clinical Outcome Scale Score 8 | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Rate of Hospitalization Through Day 28
Description: The analysis of this endpoint was performed on the intention-to-treat (ITT) population. The percentage of patients who were hospitalized was compared using a binary logistic regression analysis. The model included only the treatment group. The results were presented as odds ratios, with associated 80% CIs and p-value.
Time Frame: Day 1 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
Participants
  Yes, hospitalized | 2 | 4 | 3 | 1
  No, not hospitalized | 51 | 51 | 45 | 51
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Regression, Logistic

11. Secondary Outcome: Rate of Progression to Oxygen Therapy Through Day 28
Description: The analysis of this endpoint was performed on the intention-to-treat (ITT) population. The number and percentage of patients who progressed to oxygen therapy was presented. The percentage of patients who had progressed to oxygen therapy was compared using a binary logistic regression analysis. The model included only the treatment group. The results were presented as odds ratios, with associated 80% confidence intervals (CIs) and p-value.
Time Frame: Day 1 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
Participants
  Yes, progressed to oxygen therapy | 1 | 4 | 2 | 1
  No, did not progress to oxygen therapy | 52 | 51 | 46 | 51
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Regression, Logistic

12. Secondary Outcome: Type of Oxygen Therapy Received Through Day 28
Description: The analysis of this endpoint was performed on the intention-to-treat (ITT) population and only on those who received oxygen therapy. The number and percentage of patients who received different types of oxygen therapy was presented using descriptive statistics.
Time Frame: Day 1 to Day 28
Population: The type of oxygen therapy received was measured for all participants in the intent-to-treat (ITT) population; however, the data presented here reflects an analysis performed only on those subjects from the ITT population who received oxygen therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 1 | 4 | 2 | 1
Participants
  Supplemental oxygen | 1 | 4 | 1 | 1
  Mechanical ventilation | 0 | 0 | 1 | 0

13. Secondary Outcome: Duration of Hospitalization
Description: The duration of hospitalization was performed on the intention-to-treat (ITT) population in subjects who were hospitalized. Duration of hospitalization was summarized by treatment group using descriptive statistics (N, mean, median, standard deviation, Q1, Q3, minimum, and maximum). An ANOVA model was performed to analyze the difference between treatment groups. The model included only the treatment group. Contrasts under this model allowed for the comparisons across treatment groups. The results were presented as mean treatment difference with associated 80% confidence interval (CI) and p-value.
Time Frame: Day 1 through Day 28
Population: The duration of hospitalization was measured for all participants in the intent-to-treat (ITT) population; however, the mean length of hospitalization for each arm presented here reflects an analysis performed on only the hospitalized subjects from the ITT population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 2 | 4 | 3 | 1
days | 3.0 (0.0) | 5.75 (5.19) | 8.67 (12.42) | 3.0 (0)
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, ANOVA

14. Secondary Outcome: Mortality Rate by Day 28
Description: The analysis of this endpoint was performed on the intention-to-treat (ITT) population. The number and percentage of patients who died was presented. The percentage of patients who died was compared using a binary logistic regression. The model included only the treatment group. Contrasts under this model allowed for the comparisons across treatment groups. The results were presented as odds ratios, with associated 80% CIs and p-values.
Time Frame: Day 1 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
Number analyzed (Participants) | 53 | 55 | 48 | 52
Participants
  No, did not die | 53 | 55 | 47 | 52
  Yes, died | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Placebo Tablets vs 900 mg Dose vs 1800 mg Dose vs 3600 mg Dose; Test type: Superiority; p = 0.2, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected for approximately 1 month. All subjects were closely monitored for adverse events from informed consent for at least 18 days after the final dose of study treatment (until Day 28 ±2). Subjects who withdrew early from the study had follow-up phone calls to collect safety data until End of Study on Day 28±2.
Description: Adverse events (AE) data were collected and analyzed only for subjects who were enrolled and took at least 1 dose of study medication.
Arm/Group | Placebo Tablets | 900 mg Dose | 1800 mg Dose | 3600 mg Dose
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55 | 1/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/53 | 4/55 | 4/48 | 1/52
Other Adverse Events (participants affected / at risk) | 29/53 | 27/55 | 33/48 | 46/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Tablets (N=53) | 900 mg Dose (N=55) | 1800 mg Dose (N=48) | 3600 mg Dose (N=52)
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0
Rash maculopapular (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Tablets (N=53) | 900 mg Dose (N=55) | 1800 mg Dose (N=48) | 3600 mg Dose (N=52)
Diarrhea (Gastrointestinal disorders) | 10 | 14 | 14 | 30
Feces soft (Gastrointestinal disorders) | 2 | 1 | 4 | 2
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 4 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 5 | 6 | 6 | 12
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 1
Laboratory test abnormal (Investigations) | 7 | 5 | 5 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 5 | 3

LIMITATIONS AND CAVEATS:
Small sample size, remote study, and patients were self-sampling for the polymerase chain reaction (PCR) testing albeit under supervision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT04676867/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04676867/SAP_001.pdf